CLINICAL TRIAL: NCT02277613
Title: A Phase 2 Prospective, Randomized, Double-blind, Sham-controlled, Parallel-group, Multi-center Trial of AMI MultiStem® Therapy in Subjects With Non-ST Elevation Acute Myocardial Infarction
Brief Title: A Phase 2 Trial of AMI MultiStem® Therapy in Subjects With Non-ST Elevation Acute Myocardial Infarction
Acronym: MI-NSTEMI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B02-02; 1R44HL117572-01A1 (NIH)
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Heart Attack; NSTEMI
Keywords: stem cells
MeSH Terms: conditions — Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AMI MultiStem cells (Experimental): AMI MultiStem cells is a cell therapy medicinal product originating from adherent stem cells taken from the bone marrow of a non-related donor and expanded ex vivo.
  Interventions: Biological: AMI MultiStem cells
- Sham (Sham Comparator): Sham procedure using Micro-Infusion Catheter in coronary artery without injection.
  Interventions: Other: Sham

INTERVENTIONS:
Biological: AMI MultiStem cells — AMI MultiStem cells administration in coronary artery with a micro-infusion catheter.
  Arms: AMI MultiStem cells
Other: Sham — Sham procedure using Micro-Infusion Catheter in coronary artery without injection.
  Arms: Sham

SUMMARY:
This is a double-blind, sham-controlled clinical study to evaluate the safety and feasibility of AMI MultiStem therapy in subjects who have had a heart attack (Non-ST elevation MI).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender, 18-85 years of age, inclusive
* Diagnosis of non-ST elevation myocardial infarction (NSTEMI)
* Left Ventricular Ejection Fraction (LVEF) between ≥ 25 and ≤ 45%

Exclusion Criteria:

* Previous Coronary Artery Bypass Graft (CABG)
* Previous autologous, allogeneic bone marrow or peripheral stem cell transplant
* Previous solid organ transplant
* Anticipated need for additional planned coronary revascularization procedure(s)
* Hemodynamic instability
* Mechanical complications of the index acute myocardial infarction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 30 days
  To compare the difference in the incidence and severity of adverse events between AMI MultiStem therapy treated subjects and Sham treated subjects
To assess the effects of AMI MultiStem therapy on cardiac function | Day 120
  To compare the changes in cardiac function assessed by cardiac MRI between AMI MultiStem therapy treated subjects and Sham treated subjects

SECONDARY OUTCOMES:
To assess the effects of AMI MultiStem therapy on cardiac function | Day 365
  To compare the changes in cardiac function assessed by cardiac MRI between AMI MultiStem therapy treated subjects and Sham treated subjects
To assess the incidence of Major Adverse Cardiovascular Events (MACE) | Day 365
  To compare the incidence of MACE between AMI MultiStem therapy treated subjects and Sham treated subjects
Incidence and severity of adverse events | Day 365
  To compare the difference in the incidence and severity of adverse events between AMI MultiStem therapy treated subjects and Sham treated subjects

CONTACTS AND LOCATIONS:
Overall Officials: Marc Penn, MD, Principal Investigator — Summa Health System
Locations (11):
- United States (11):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Los Angeles, California
  - Clearwater, Florida
  - Gainesville, Florida
  - Tampa, Florida
  - Detroit, Michigan
  - Akron, Ohio
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah
  - Madison, Wisconsin